CLINICAL TRIAL: NCT06660355
Title: Phase II Randomized Study of Ruxolitinib vs Prednisone as First-Line Therapy for Chronic Graft vs Host Disease Needing Systemic Therapy
Brief Title: Ruxolitinib vs Prednisone as First-line Therapy for cGVHD Needing Systemic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23051
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft-versus-host Disease (cGVHD)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib Treatment Arm (Experimental): Ruxolitinib is administered as 10 mg orally twice daily in 28-day cycles.
  Interventions: Drug: Ruxolitinib
- Prednisone Treatment Arm (Active Comparator): Prednisone will be started at 1mg/kg/day based on patient current body weight in kilograms.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is a Janus kinase inhibitor.
  Arms: Ruxolitinib Treatment Arm
Drug: Prednisone — Prednisone is a glucocorticoid.
  Arms: Prednisone Treatment Arm

SUMMARY:
Allogeneic transplant is potentially curative for hematological malignancies but its use is limited by the development of GVHD. Ruxolitinib now has FDA approval for treatment of chronic GVHD that has failed 1-2 prior lines of therapy based on a prior large, randomized phase III study. Given this evidence of safety and efficacy in the early refractory setting (after prednisone failure), Ruxolitinib represents an ideal agent to test in the primary therapy setting. Here investigators propose a phase 2 randomized study to compare Ruxolitinib to prednisone as a first-line therapy in the treatment of chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Karnofsky performance status ≥60%.
* Patients with a diagnosis of chronic GVHD per NIH diagnostic criteria5 who are in need for first systemic therapy as per treating physician's discretion, Overlap chronic GVHD will be allowed.
* No new immune suppressive therapy added within preceding 2 weeks prior to study enrolment.
* Able to take oral medications.
* Participants must have adequate organ and marrow function as defined below:

  1. absolute neutrophil count ≥1,000/mcL
  2. platelets ≥30,000/mcL
  3. Hemoglobin ≥ 7 g/dL
  4. Bilirubin ≤ 3 times institutional upper limit of normal (ULN) unless attributable to GVH

  d. AST(SGOT)/ALT(SGPT) ≤5 × institutional ULN unless attributable to GVH e. creatinine clearance ≥30 ml/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study drug administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Previously treated with systemic immune suppressive therapy for chronic GVHD (where the indication for start of that systemic immune suppressive therapy was chronic GVHD).
* Patients with clinically significant or uncontrolled cardiovascular disease, including unstable angina, acute myocardial infarction, or stroke within 6 months, New York Heart Association class III or IV heart failure will be excluded.
* Relapse malignancy post- transplant.
* Active hepatitis B, hepatitis C and HIV will be excluded.
* Any uncontrolled infection at the time if enrollment will be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Ruxolitinib.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and lactating women are excluded from this study because of the potential for teratogenic or abortifacient effects and an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Ruxolitinib, breastfeeding should be discontinued if the mother is treated with Ruxolitinib.
* Current or history of active Tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | 6 months
  Treatment Success is defined as C7D1 NIH CR/PR without death or new line of immune suppressive therapy and will be estimated for both arms.

SECONDARY OUTCOMES:
Treatment Success Rate | 6 months
  The proportion of subjects who are alive with NIH CR/PR, no new systemic therapy for cGVHD, and < 0.25 mg/kg/day prednisone at C7D1 with 95% CI for each arm will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Khimani, MD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - Univ of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Virginia Commonwealth University, Richmond, Virginia